CLINICAL TRIAL: NCT00956891
Title: Therapeutic Effects Including Short-term Changes And Long-term Outcomes of Liver Failure Patients Caused by Chronic Hepatitis B After Single Transplantation With Autologous Bone Marrow Mesenchymal Stem Cells.
Brief Title: Therapeutic Effects of Liver Failure Patients Caused by Chronic Hepatitis B After Autologous MSCs Transplantation
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: The Third Affliated Hospital of Sun Yat-sen University, The Third Affliated Hospital of Sun Yat-sen University
Other Study IDs: SunYat-senU 5010 hepatitisB
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2009-08

CONDITIONS: Liver Failure; Mesenchymal Stem Cells
Keywords: short-term effects; long-term follow-up; liver failure patients; autologous MSCs transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group A: autologous MSCs transplantation were performed plus medical treatments (reducibility glutathione, glycyrrhizin, ademetionine, polyene phosphatidylcholine, alprostadil, and human serum albumin)
- group B: only medical treatments (reducibility glutathione, glycyrrhizin, ademetionine, polyene phosphatidylcholine, alprostadil, and human serum albumin) were performed without autologous MSCs transplantation.

SUMMARY:
The study aimed to investigate the short-term efficacy and long-term prognosis of liver failure patients caused by hepatitis B after single transplantation with autologous marrow mesenchymal stem cells (MMSCs). Liver failure inpatients caused by hepatitis B were recruited and received the same medical treatments, among whom some patients underwent single transplantation with autologous MMSCs and other patients with matched age, gender and biochemical indexes [alanine aminotransferase (ALT), albumin (ALB), total bilirubin (TBIL), prothrombin time (PT) and Model for End-stage Liver Disease (MELD) ] were in control group. A total of 120 ml bone marrow were obtained from patients, diluted and separated. Then MMSCs suspension were slowly transfused into the liver through the proper hepatic artery by interventional procedures. The levels of ALB, TBIL, PT and MELD score of patients in translation group were compared with those in control group. In 3 ~ 48 months of follow-up, differences in long-term outcomes such as incidence of HCC (hepatocellular carcinoma) and mortality between two groups were compared.

DETAILED DESCRIPTION:
A total of 527 patients with chronic hepatitis B induced liver failure were recruited from May 2005 to June 2009 from our department. The diagnoses of chronic hepatitis B and liver failure were based on previously described criteria. All patients received the same medical treatments (reducibility glutathione, glycyrrhizin, ademetionine, polyene phosphatidylcholine, alprostadil, and human serum albumin). Informed consent was obtained before study. Among these patients, 53 received transplantation with autologous MMSCs. The day of surgery served as the first day of observation. And 105 patients with matched age, gender and some biochemical indexes (ALT, ALB, TBIL, PT and MELD ) were served as controls.

ELIGIBILITY:
Inclusion Criteria:

* Liver failure

Exclusion Criteria:

* HBV negative

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver failure patients with HBV infection
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2005-05; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Short-term therapeutic effects of transplantation. | 1 to 4 weeks after transplantation
  Biochemical indexes [alanine aminotransferase (ALT), albumin (ALB), total bilirubin (TBIL), prothrombin time (PT) and Model for End-stage Liver Disease (MELD) ] were compared 1 to 4 weeks after transplantation.

SECONDARY OUTCOMES:
Long-term outcomes of transplantation. | 3 ~ 48 months years after transplantation
  In 3 ~ 48 months of follow-up, incidence of HCC (hepatocellular carcinoma) and mortality were compared between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-liang Gao, Dr, Study Director — Department of Infectious Diseases, 3rd Affiliated Hospital of Sun Yat-sen University, China
Locations (1):
- The Third Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong, China